CLINICAL TRIAL: NCT01845415
Title: A Community-Based Intervention to Prevent Fall Injuries to Young Children in the Home
Brief Title: Intervention to Prevent Fall Injuries to Young Children in the Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Barbara A. Morrongiello, PhD, C. Psych., Professor, University of Guelph
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 13AP011; 450083 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Social Marketting Only (Active Comparator): Two communities receive a social marketing campaign to reduce child falls in the home.
  Interventions: Behavioral: Social Marketing Campaign
- No treatment Control (No Intervention): two communities receive no intervention
- Social Marketing plus Intervention (Active Comparator): Two communities receive the social marketing campaign and additional intervention components
  Interventions: Behavioral: Social Marketing Campaign; Behavioral: Intervention components

INTERVENTIONS:
Behavioral: Social Marketing Campaign — The campaign will involve distribution of posters throughout the communities promoting awareness of the consequences of fall injuries and encouraging people to go to an website that provides safety information and injury stories.
  Arms: Social Marketing plus Intervention; Social Marketting Only
Behavioral: Intervention components — Doctors and nurses in these communities will perform health education to parents of 1 through 4 year olds around the risks of falls in the home when these parents visit the doctor for regular visits. Also, several parenting classes in these communities will be modified to include educational videos and discussion of these issues
  Arms: Social Marketing plus Intervention

SUMMARY:
Currently, six Public Health Units (PHUs) in Southwestern Ontario are taking part in the developed and implementation of a social marketing intervention campaign aimed at lowering the incidence of falls to children in the home; City of Hamilton - Public Health Services (Control), Durham Public Health, Haldimand-Norfolk Health Unit, Niagara Region Public Health, Wellington-Dufferin-Guelph Public Health and Windsor Public Health (Control). This campaign is based on community-based intervention research and 'best practices' for improving parent attitudes and behaviours toward child safety. The campaign will focus on increasing parents' awareness and knowledge of fall injuries, positively impact parental attitudes to motivate them to want to implement strategies to reduce fall risks, and increase parental safety practices that would counteract the most common mechanisms that contribute to home falls for children at these young ages. The campaign will run from September 2013 through August 2014. The PHUs' social marketing campaign will strategically disseminate different materials to their respective communities: printed materials (posters, pamphlets), video modules about parenting safety, safety information through an e-Health website, and direction communication with parents through Family Health Team practitioners.

The proposed research project will request archival data from Canadian Institute of Health Information (CIHI), specifically from their National Ambulatory Care Reporting System (NACRS), on frequency of falls in the home to determine the extent to which the social marketing campaign is effective. Comparing pre-, during and post-intervention levels in the PHU communities will determine if and which social marketing strategies were effective. Additionally, random digit dialing will be used to assess pre vs post parental fall related attitudes, behaviors and intervention exposure. This evaluation will provide the first ever test of a community level intervention to reduce childhood falls in the home in Canada and will provide valuable information about what constitutes 'best practices' for preventing falls in the home among children 1 through 4 years of age.

ELIGIBILITY:
Inclusion Criteria:

* must be a parent or primary care giver of a child 1 through 4 years of age
* must live in one of the designated communities (by postal code)

Exclusion Criteria:

-

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Emergency Department Visits due to Falls in the Home from pre- to post- intervention periods | One year pre intervention (Oct. 2012- Oct 213), one year post intervention (Oct 2014-Oct 2015)
  We will be comparing the rate of injury due to falls in the home during the pre-intervention period with that during the post-intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guelph, Guelph, Ontario, Canada